CLINICAL TRIAL: NCT03949946
Title: Is Lipid Composition Mapping Using Magnetic Resonance Imaging an Effective Early Detection Tool for Breast Cancer in High Risk Populations?
Brief Title: Is Lipid Mapping an Effective Early Detection Tool for Breast Cancer in High-risk Populations?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-025-19
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: lipid composition; MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk: Female participants confirmed to be BRCA1/2 or TP53 gene carriers
  Interventions: Procedure: Magnetic resonance imaging (MRI)
- Patients: Female participants confirmed to have invasive ductal carcinoma of the breast
  Interventions: Procedure: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic resonance imaging (MRI) — MRI scan uses radio waves in a magnetic field to obtain images of the breast. It is non-invasive and participants will not be exposed to harmful radiation. An image contrast agent will be used to enhance image clarity. Participants will be scanned lying face-down on a specially-designed bed and ear protectors will be provided to screen out background noise.

SUMMARY:
This study aims to investigate if lipid composition mapping using magnetic resonance imaging could improve early and accurate cancer detection in genetic mutation carriers at high risk of breast cancer. It is hypothesised that there is a significant difference in the extent of spatial variation in lipid composition in breast from MRI between genetic mutation carriers and patients with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a major and expanding societal challenge despite the significant improvement in survival rate. The current screening method has been shown to lead to overtreatment, prompting the development of accurate early detection approaches targeting underlying clinical features. Patients with BRCA1/2 and TP53 genes are at risk of breast cancer and receive annual surveillance. However, the current diagnostic approach relies on detecting the changes to the growth of tumour only once cancer is well under development. Detecting earlier changes to breast fatty tissue may detect patients earlier and more accurately.

Breast fatty tissue is composed of different fatty acids and a difference in the fatty acid composition has been shown in BRCA1/2 gene carriers. Measurement of lipid composition can be achieved using a specialist magnetic resonance spectroscopy method, but is limited to sampling a small area and is unable to provide the full picture of lipid composition distribution during early cancer growth. Recently, magnetic resonance chemical shift imaging, through combining magnetic resonance spectroscopy and imaging approaches, has been developed to provide lipid composition maps of the entire breast.

The investigators propose to perform lipid mapping in the breasts of 20 genetic mutation carriers at high risk of breast cancer and 20 patients with newly diagnosed breast cancer to examine the sensitivity of the method. The overarching aim is to improve early and accurate cancer detection in genetic mutation carriers at high risk of breast cancer through the assessment of whole breast lipid composition.

ELIGIBILITY:
Inclusion Criteria:

* female over 18 years old
* BRCA1/2 or TP53 gene carriers (high-risk group)
* invasive ductal carcinoma of the breast (patient group)
* not having any metabolic disorders (e.g., diabetes)
* not on any long term medications that may affect lipid metabolism (e.g., statins)

Exclusion Criteria:

* female under 18 years old
* male
* affected by metabolic disorders (e.g., diabetes)
* on long term medications that affect lipid metabolism (e.g., statins)
* contraindicated for MR investigations (poor renal function and metal implants)
* concurrent cancer in other sites
* concurrent hormone treatment, chemotherapy or underwent surgery
* non-English speakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female participants confirmed to be BRCA1/2 and TP53 gene carriers and females participants confirmed to have invasive ductal carcinoma of the breast.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Saturated fatty acids in breasts of patients and high-risk group | Baseline
  Saturated fatty acids (SFA) from tumour border and fatty tissue in patients and fibroglandular and fatty tissue in high-risk group
  SFA will be measured in percentage (%)
Monounsaturated fatty acids in breasts of patients and high-risk group | Baseline
  Monounsaturated fatty acids (MUFA) from tumour border and fatty tissue in patients and fibroglandular and fatty tissue in high-risk group
  MUFA will be measured in percentage (%)
Polyunsaturated fatty acids in breasts of patients and high-risk group | Baseline
  Polyunsaturated fatty acids (PUFA) from tumour border and fatty tissue in patients and fibroglandular and fatty tissue in high-risk group
  PUFA will be measured in percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Jiabao He, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Biomedical Imaging Centre, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No